CLINICAL TRIAL: NCT05068596
Title: Influence of Loaded Functional Strength Training From a Plantigrade Foot Position Using Shoe Holder on Hip and Knee Extensors Strength and Function Walking Capacity in Children With Spastic Hemiplegic Cerebral Palsy
Brief Title: Effect of Loaded Functional Training on Hemiplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, hanaa mohsen, lecturer in the department of paediatrics and paediatric surgery , faculty of physical therapy, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hana 9
Record Dates: First submitted 2021-09-12; First posted 2021-10-06 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-02

CONDITIONS: Hemiplegic Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study groip (Experimental): received the designed physical therapy program as the control group. In addition, they received progressive resistive functional strength training in the plantigrade foot position.
  Interventions: Other: expermintal
- control group (Other): received a designed physical therapy program
  Interventions: Other: CONTROL

INTERVENTIONS:
Other: expermintal — progressive resistive functional strength training in the plantigrade foot position plus designed physical therapy program
  Arms: study groip
Other: CONTROL — Designed physical therapy program
  Arms: control group

SUMMARY:
weakness of lower limb is common in cp children

ELIGIBILITY:
Inclusion Criteria:

* age 10-12
* level I,II according to GMFCM
* Able to follow and understand instructions

Exclusion Criteria:

* visual and respiratory disorder

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Muscle strength dynamometry | pre and post three month of intervention high score indicate improvement
  The gold standard for evaluating isometric muscle strength is the portable dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa M Abd-Elfattah, ph.d, Principal Investigator — lecturer
Locations (1):
- Hanaa Mohsen Abd-Elfattah, Cairo, Egypt